CLINICAL TRIAL: NCT00477620
Title: Study of Myopia Acquisition and Prevention in a Randomised Trial
Brief Title: Study of Myopia Acquisition and Prevention
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FR-2005-01-01
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2009-02-23 (Estimated); Status verified 2009-02

CONDITIONS: Myopia
Keywords: Myopia; Prevention
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Wearing of reading glasses during prolonged near work

SUMMARY:
Purpose:

To determine whether the use of reading glasses blocks the near work mediated increased incidence of myopia in healthy school children.

Methods:

SMART enrolled 115 emmetropic children (ages 7-9 years). The children were recruited in the Principality of Liechtenstein. They were randomly assigned to either the control group (n=52) or to receive reading glasses with a lens power of +2.0 dioptres (n=63). The primary outcome measure was progression towards myopia as determined by autorefraction after cycloplegia. The secondary outcome measure was change in biometry measurements of corneal curvature, axial length, anterior chamber depth, crystalline lens thickness, and vitreous chamber depth using partial coherence interferometry.

ELIGIBILITY:
Inclusion Criteria:

* Emmetropia

Exclusion Criteria:

* Ametropia

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2004-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexaner Reis, PD Dr. med., Study Chair — Augenwerk Liechtenstein